CLINICAL TRIAL: NCT06311773
Title: Pivotal Multicenter Trial of the Boomerang® Catheter for Percutaneous Deep Vein Arterialization (pDVA)
Brief Title: Pivotal Trial of the Boomerang Catheter for pDVA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aveera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol # 24-01
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treated with Boomerang Catheter (Experimental)
  Interventions: Device: Boomerang Catheter

INTERVENTIONS:
Device: Boomerang Catheter — The study device used for this procedure makes an anastomosis between a tibial vein and a tibial artery to direct blood flow around blocked arteries.

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of the Boomerang Catheter for percutaneous Deep Venous Arterialization (pDVA) to treat no-option Chronic Limb-Threatening Ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age ≥ 18 years
2. Patient has confirmed clinical diagnosis of Rutherford Category (RC) 5 or 6 Chronic Limb-Threatening Ischemia (CLTI) with previous angiogram or hemodynamic evidence (e.g., ABI ≤ 0.39, TP / TcPO2 < 30 mm Hg) demonstrating severely diminished arterial perfusion of the index limb.
3. Assessment by the PI and an Independent Review Committee (IRC) determines that patient has no option for conventional distal bypass, surgical or endovascular therapy for limb salvage.
4. Inflow artery criteria:

   • Imaging confirmation of patent inflow artery (< 50% stenosis) from Aortic bifurcation to tibial trifurcation.
5. Target conduit vein criteria:

   • Duplex ultrasound confirms that vein is free from thrombus, contiguous from the intended anastomosis site through the lateral plantar vein, and ≥ 2.0mm lumen-lumen diameter (with tourniquet applied) throughout.
6. Patient may be scheduled for a planned minor amputation (toe, ray, or trans-metatarsal) within 30 days after index procedure.
7. Prior stent(s) to inflow arteries (i.e., Iliac, SFA, Popliteal) are allowed.
8. Patient is willing and able to provide written informed consent.
9. Patient meets institutional criteria for procedure clearance and is able to comply with study requirements per PI judgement.
10. Diabetic patients have adequate glycemic control per investigator judgement.
11. Female patients of childbearing potential have a negative pregnancy test within 7 days prior to index procedure (urine)
12. Patient is enrolled in a wound care network and has an adequate support network to ensure compliance with medication regimen and follow-up study visits.
13. PI determines that the primary wound is stable (e.g., not rapidly deteriorating or showing signs of healing).

Exclusion Criteria:

1. Life expectancy < 12 months.
2. Patient has a lower extremity vascular disease that may inhibit the procedure and/or jeopardize wound healing (e.g., vasculitis, Buerger's disease, significant edema in the target limb, deep venous thrombus in the target vein, hyperpigmentation, or medial ulceration above the ankle).
3. Patient is dialysis dependent.
4. Significant acute or chronic kidney disease with a serum creatinine of > 2.5 mg/dl in patients not undergoing dialysis.
5. Prior peripheral arterial bypass procedure on index limb within 30 days.
6. Previous major amputation of the target limb or absence of adequate viable tissue for below-ankle (e.g., mid-foot) amputation.
7. Patient is non-ambulatory due to above-ankle amputation of contralateral limb.
8. The patient is currently participating in another investigational drug or device study that has not completed the primary endpoint and that clinically interferes with the endpoints of this study per PI judgement.
9. Patient has known hypersensitivity or contraindication to materials used during the procedure (cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers) or a known contrast sensitivity that cannot be adequately pre-medicated.
10. Patient cannot be adequately treated with study medications due to known contraindication to aspirin, ADP antagonists such clopidogrel, prasugrel or ticagrelor, or anticoagulants such as heparin or bivalirudin.
11. Patient has had a stroke within the previous 3 months with residual Rankin score of ≥ 2.
12. NYHA Class IV heart failure which may compromise patient's ability to safely undergo a percutaneous procedure, per PI judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Amputation Free Survival (AFS) | 6-months
  Freedom from above-ankle amputation of the index limb or death (any cause) at 6 months, compared to a literature derived performance goal.

SECONDARY OUTCOMES:
Technical success | During index procedure
  Successful deployment of the Boomerang Catheter to the anastomosis site, creation of an anastomosis, and confirmation of fistula flow using angiography or Doppler ultrasound immediately post catheter activation.
Procedural success | Immediately post index procedure
  confirmation of retrograde fistula flow in the target tibial vein conduit at index procedure completion.
Limb salvage | 3 years post index procedure
  Freedom from above-ankle amputation of the index limb.
Primary patency | 1 year post index procedure
  Time from fistula creation to the first intervention to maintain or reestablish flow through the fistula or to fistula occlusion.
Primary assisted patency | 1 year post index procedure
  Time from fistula creation to the first occlusion of the fistula.
Secondary patency | 1 year post index procedure
  Time from fistula creation to abandonment (e.g., decision to decline intervention due to occlusion) of the fistula.
Target wound healing | 1, 3, 6, 9-months, and 1-year
  Complete or in-process healing of the patient's target wound(s).
Complete wound healing | 1, 3, 6, 9-months, and 1-year
  Complete healing of all the patient's ischemic wound(s) in the index limb.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Olive View-UCLA Medical Center, Sylmar, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - PIH Whittier Hospital, Whittier, California
  - EndoVascular Consultants, Wilmington, Delaware
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Vascular Institute at AMI, Galloway, New Jersey
  - American Endovascular and Amputation Prevention, West Orange, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Sunrise Vascular, Murphy, North Carolina
  - Advanced Vascular Centers, Tigard, Oregon
  - Penn Medicine, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - HOPE Vascular and Podiatry, Houston, Texas
  - University of Washington Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No